CLINICAL TRIAL: NCT05281185
Title: Clinical Outcomes of Low Dose Pharmacokinetic-guided Extended Half-life FVIII Concentrates Versus Low Dose Standard Prophylaxis in Thai Severe Haemophilia A Patients
Brief Title: Clinical Outcomes of Low Dose PK-guided EHL FVIII Concentrates Versus Standard Prophylaxis in Severe Haemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PedHemophiliaCU
Record Dates: First submitted 2022-02-08; First posted 2022-03-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-01

CONDITIONS: Severe Hemophilia A Without Inhibitor
Keywords: severe hemophilia A; extended FVIII concentrates; low dose prophylaxis; MyPKFiT
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Patients aged 5-25 years with clinically severe haemophilia A (FVIII:C ≤3%), no inhibitor, on low-dose weight-based prophylaxis at King Chulalongkorn Memorial Hospital (KCMH) Thailand
Masking Description: Open label, all participants received individual low-dose PK-guided extended FVIII concentrates prophylaxis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Severe haemophilia A patients with weight-based prophylaxis (Active Comparator): Severe haemophilia A patients with low-dose standard half-life concentrates weight-based prophylaxis
  Interventions: Drug: standard half-life FVIII concentrates with weight-based dosing
- Severe haemophilia A patients with low dose extended half-life PK-guided prophylaxis (Experimental): Severe haemophilia A patients with low-dose extended half-life concentrates PK-guided prophylaxis
  Interventions: Drug: Extended half-life FVIII concentrates with PK-guided dosing

INTERVENTIONS:
Drug: Extended half-life FVIII concentrates with PK-guided dosing — Extended half-life FVIII concentrates with PK-guided dosing as low-dose factor replacement prophylaxis (10-20u/kg, 2-3 times/week) for 6 months in severe haemophilia A patients that previously receive weight-based factor replacement prophylaxis
  Arms: Severe haemophilia A patients with low dose extended half-life PK-guided prophylaxis
Drug: standard half-life FVIII concentrates with weight-based dosing — standard half-life FVIII concentrates with weight-based dosing, that current patients' regimen before enrolling in this study
  Arms: Severe haemophilia A patients with weight-based prophylaxis

SUMMARY:
Individualised pharmacokinetic (PK)-guided dosing of extended half-life (EHL) FVIII concentrates prophylaxis may reduce hemophilia A bleeding events than previous prophylactic regimen.

Methods A single-centre prospective cohort study, the investigators recruited consecutive eligible patients aged 5-25 years with clinically severe haemophilia A (FVIII:C ≤3%), no inhibitor, on low-dose weight-based prophylaxis at King Chulalongkorn Memorial Hospital (KCMH) from July 2021 to February 2022.

All of patients with clinically severe haemophilia A received low dose weight-based standard half-life FVIII concentrates replacement prophylaxis for ≥ 1 year prior to enrolment in the study.

The data of annual bleeding rate (ABR), annual joint bleeding rate (AJBR), annual FVIII use (prophylactic and breakthrough bleeding dosing) in the last 6 months before the study and number of target joints were collected at the beginning of the study.

Baseline variables, including age and weight, were recorded before performing the analyses using online medical device (www.mypkfit.com).

Wash-out period for 72 hours, each participant subsequently received a dose of 20 IU/kg FVIII by intravenous injection. Blood samples were collected and the concentration of FVIII was measured two times at 3 h and 48 h or 72 h after injection by one-stage technique. Desired FVIII trough levels were selected in this study as 1%. Individually proper regimen were selected by discussion with patients and families.

All of participant individually underwent dose calculation of EHL factor VIII concentrates and received low dose PK-guided regimen (10-20u/kg, 2-3times/week) with EHL FVIII concentrates for 6 months. If breakthrough bleeding occurs, FVIII concentrates 500 U intravenous injection immediately.

ABR, AJBR, HJHS and annual FVIII concentrates use were again prospectively recorded during intervention period after PK adjustment for 6 months.

Primary objectives To compare clinical outcomes including annual bleeding rate (ABR), annual joint bleeding rate (AJBR) and Haemophilia joint health score (HJHS) before and after switching from standard half-life (SHL) to Extended half-life (EHL) factor VIII concentrates with adjusted dosing by PK-guided program (MyPKFiT®) in severe haemophilia A patients Secondary objectives To compare factor VIII concentrates consumption before and after using PK-guided program (MyPKFiT®) adjusting dose of factor VIII infusion in severe HA patients.

DETAILED DESCRIPTION:
Clinical Outcomes of Low Dose Pharmacokinetic-guided Extended Half-life Versus Low Dose Standard Half-life FVIII Concentrates Prophylaxis in Thai Severe Haemophilia A Patients

Haemophilia A (HA) is a X-linked inherited bleeding disorders caused by a deficiency in the clotting factor VIII (FVIII). The degree of deficiency was determined by a patient's FVIII level and clinical bleeding phenotype. Clinically severe haemophilia A (FVIII < 1 IU/dL) typically present with recurrent joint and muscle bleeds. They may also experience spontaneous and potentially fatal bleeds in any tissue.

The standard of care for all patients with severe haemophilia A is regular factor replacement prophylaxis with clotting factor concentrates or other homeostasis products to maintain homeostasis for preventing bleeding, especially joint haemorrhages, which lead to arthropathy and disability. People with haemophilia A initiated on early prophylaxis (i.e., primary or secondary prophylaxis) have shown the best long-term outcomes. Therefore, the use of prophylaxis is always recommended over episodic therapy that no longer be a long-term treatment option.

The aim of prophylaxis has been to convert a person with severe haemophilia (baseline FVIII <1 IU/dL) to a bleeding phenotype typical of moderate or mild haemophilia who seldom experienced spontaneous bleeding and had much better preservation of joint function by maintaining factor levels above 1 IU/dL (1%) at all times. However, there has been increasing recognition and evidence that factor trough levels of 1-3 IU/dL (1%-3%) are insufficient to totally prevent bleeds in all people with haemophilia and allow occasional clinical and subclinical bleeds. And when baseline FVIII:C levels are above 15 IU/dL (15%), spontaneous bleeding is uncommon, traumatic bleeding during high activity is few.

The World Federation of Haemophilia (WFH) strongly recommends that prophylaxis should be individualised, taking into consideration patient bleeding phenotype, joint status, level of physical activity, individual pharmacokinetics, compliance, and patient self-assessment and preference in severe haemophilia patients. If patients continue to experience bleeds, their prophylaxis regimen should be escalated (in dose/frequency or both) to prevent bleeding. In countries with significant healthcare constraints and for patients with limited access to clotting factor concentrates, less intensive prophylaxis should be used over episodic therapy.

By Pharmacokinetic-guided calculation, the plasma activity level of the infused factor is still above the level considered critical to prevent bleeding. This critical threshold is often assumed to be 0.01-0.03 IU/mL although different thresholds have been proposed for differing levels of physical activity or tendency to bleed.

An old full PK study for haemophilia A patients requires a washout period of 72 h and sample collection for a total of 10 time-points after the infusion of the coagulation factor. In the recent years, population-based PK (PopPK) application was developed, myPKFiT®, obtained using just at least two sampling points that support optimal use of recombinant factor VIII (rFVIII) (Advate®; Shire plc, Dublin, Ireland) for treatment of haemophilia patients.

Based on pharmacokinetics (PK), increasing infusion frequency will result in reduced FVIII consumption and a more stable factor level although it may have a negative impact on adherence. In many countries, extended half-life (EHL) FVIII concentrates play role in severe haemophilia A because of median 1.3-1.6-fold extension in half-life reducing their dosing frequency from 3- to 2-times weekly. A major aim of most modifications was to facilitate improved pharmacokinetics (PK) that allow a patient to dose less frequently than with standard half-life factor products and positive impact on adherence.

Prophylaxis should enable people with haemophilia to lead healthy and active lives including participation in most physical and social activities (at home, school, work, and in the community), similar to the non-haemophiliac population.

Methods In this single-centre prospective cohort study, we recruited consecutive eligible patients aged 5-25 years with clinically severe haemophilia A (FVIII:C ≤3%) at King Chulalongkorn Memorial Hospital (KCMH) from July 2021 to February 2022. Participants were recruited through their annual clinic visit or by a letter of invitation. The study was approved by Institutional Review Board (IRB) Human Research, research affairs, faculty of medicine, Chulalongkorn university, Thailand (Certificate 222/64). Informed consent was obtained according to the Declaration of IRB Human Research, research affairs, faculty of medicine, Chulalongkorn university, Thailand.

Inclusion/exclusion criteria The inclusion criteria were as follows: (1) severe or moderate with clinically HA with a baseline FVIII level of ≤3 IU/dL, (2) age 5-25 years, (3) > 50 exposure days (EDs) without inhibitor, (4) close proximity to the comprehensive care center at KCMH, (5) compliant to treatment, and (6) use of the pre-study prophylaxis regimen for ≥ 1 year prior to enrolment in the study.

The exclusion criteria were as follows: (1) history of FVIII inhibitor (titer > 0.6 Bethesda units [BU]) and detectable FVIII inhibitor at screening (titer > 0.6 BU), and (2) planned major surgery, and (3) concomitant serious conditions including symptomatic human immunodeficiency virus (HIV) infection, juvenile rheumatoid arthritis, metabolic bone disease, or other conditions known to mimic or cause joint diseases.

2.1 | Procedures and variables All of patients with clinically severe haemophilia A received low dose weight-based standard half-life FVIII concentrates replacement prophylaxis for ≥ 1 year prior to enrolment in the study. The data of annual bleeding rate (ABR), annual joint bleeding rate (AJBR), annual FVIII use (prophylactic and breakthrough bleeding dosing) in the last 6 months before the study and number of target joints were collected at the beginning of the study.

The annual bleeding rate (ABR) and annual joint bleeding rate (AJBR) were collected by strictly bleeding recorded events from each patients with presenting to doctor in every haemophilia clinic visit.

Target joints were defined according to the World Federation of Haemophilia 2020 guidelines. Joint status was assessed using Haemophilia joint health score (HJHS) and clinical assessment for all patients.

The annual factor consumption was collected by strictly recorded by the patients including prophylaxis and breakthrough bleeding dosing with presenting to doctor in every haemophilia clinic visit.

Baseline variables, including age and weight, were recorded before performing the analyses using online medical device (www.mypkfit.com). The calculation in myPKFiT® is based on clinical study data from a published population PK model using Advate® (standard half-life FVIII concentrates) and Adynovate® (extended half-life FVIII concentrates) of Takeda Ltd. The PK model was integrated with a Bayesian algorithm and uses a 2-compartment model to display an estimated individual curve of FVIII over time. These estimated PK parameters are used to provide dose guidance to maintain a desired FVIII activity level throughout the chosen dose interval.

Following a bleed-free period of two weeks before the baseline assessment, patients did not undergo FVIII infusion for at least 72 h prior to estimate of PK parameters initiation. Each participant subsequently received a dose of 20 IU/kg FVIII by intravenous injection. Blood samples were collected and the concentration of FVIII was measured two times at 3 h and 48 h or 72 h after injection by one-stage technique. The output provided by myPKFiT® included FVIII half-life, clearance, volume of distribution at steady state and hours until trough level. Desired FVIII trough levels were selected in this study as 1%. Regimen selection (frequency every 72/96 hr and infusion day) took into account time to trough level and the simulated levels shown at different times, checked against the periods the patient needed to be better protected, according to his activities.

All of participant individually underwent dose calculation of EHL factor VIII concentrates and received low dose PK-guided regimen (10-20u/kg, 2-3times/week) with EHL FVIII concentrates for 6 months. If breakthrough bleeding occurs, FVIII concentrates 500 U intravenous injection immediately and closely observe if bleeding or symptoms persists, another dose of FVIII concentrates is indicated in the next 12 hours.

During the study, patients followed up in haemophilia clinic every months for history taking, physical examination and presenting record of bleeding events and factor consumption.

ABR, AJBR, HJHS and annual FVIII concentrates use were again prospectively recorded during intervention period after PK adjustment for 6 months. Haemarthrosis was first suspected by the patient, based on location, and confirmed by the haematologist at the visit according to his/her clinical judgement after physical/clinical examination.

For further subgroup analysis, patients were categorised into groups according to

1. Their age (older or younger than 15 years), because of differences in pharmacokinetics related to age and body weight, the generally healthier joints in younger patients
2. Their target joints (target joints or no target joints), the patients had target joints more risk of spontaneous bleeding and required high though level more than no target joint group

2.2 | Statistical analysis Data are summarised as median and interquartile range (percentile 25-percentile 75) for continuous variables, and frequency and percentage for discrete variables. Comparison of clinical outcomes was performed with the Wilcoxon rank test for paired samples, and changes in FVIII consumption were analysed using the Student t test for paired samples, after confirming the criteria for using parametric methods. Significance level was set at P < .05.

Primary objectives To compare clinical outcomes including annual bleeding rate (ABR), annual joint bleeding rate (AJBR) and Haemophilia joint health score (HJHS) before and after switching from standard half-life (SHL) to Extended half-life (EHL) factor VIII concentrates with adjusted dosing by PK-guided program (MyPKFiT®) in severe haemophilia A patients

Secondary objectives To compare factor VIII concentrates consumption before and after using PK-guided program (MyPKFiT®) adjusting dose of factor VIII infusion in severe HA patients.

ELIGIBILITY:
Inclusion Criteria:

1. severe or moderate with clinically HA with a baseline FVIII level of ≤3 IU/dL
2. age 5-25 years
3. > 50 exposure days (EDs) without inhibitor
4. close proximity to the comprehensive care center at KCMH
5. compliant to treatment
6. use of the pre-study prophylaxis regimen for ≥ 1 year prior to enrolment in the study.

Exclusion Criteria:

1. history of FVIII inhibitor (titer > 0.6 Bethesda units [BU]) and detectable FVIII inhibitor at screening (titer > 0.6 BU)
2. planned major surgery, and (3) concomitant serious conditions including symptomatic human immunodeficiency virus (HIV) infection, juvenile rheumatoid arthritis, metabolic bone disease, or other conditions known to mimic or cause joint diseases.

Ages: 5 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Haemophilia A (HA) is a X-linked recessive bleeding disorders, so only male patients effected this disease.
Enrollment: 15 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changing bleeding rate after switch from SHL to EHL with PK-guided dosing | 6 months
  To compare bleeding events including annual bleeding rate (ABR) in numbers per year, and annual joint bleeding rate (AJBR) in numbers per year before and after switching from standard half-life (SHL) to Extended half-life (EHL) factor VIII concentrates with adjusted dosing by PK-guided program (MyPKFiT®) in severe haemophilia A patients The higher scores mean the worse outcome.
Changing the joints health outcomes after switch from SHL to EHL with PK-guided dosing | 6 months
  Haemophilia joint health score (HJHS) version 2.1 before and after switching from standard half-life (SHL) to Extended half-life (EHL) factor VIII concentrates with adjusted dosing by PK-guided program (MyPKFiT®) in severe haemophilia A patients Haemophilia joint health score (HJHS) assessed by physical examination of joint health including length of motion, swelling, pain and pattern of gait.
  The higher scores mean the worse outcome. The minimal score is zero and the maximal score is 178.

SECONDARY OUTCOMES:
Changing factor consumption after using PK-guided program | 6 months
  To compare annualised factor VIII concentrates consumption in units of factor per year before and after using PK-guided program (MyPKFiT®) adjusting dose of factor VIII infusion in severe HA patients.
  The annual factor consumption of previous study period was collected by strictly recorded by the patients including prophylaxis and breakthrough bleeding dosing with presenting to doctor in every haemophilia clinic visit during receiving SHL prophylaxis.
  During the study, patients followed up in haemophilia clinic every months for history taking, physical examination and presenting record of bleeding events and factor consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric department, Faculty of medicine, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April-June 2022

REFERENCES:
- [Derived] Rakmanotham A, Moonla C, Sosothikul D. Clinical outcomes of low-dose pharmacokinetic-guided extended half-life versus low-dose standard half-life factor VIII concentrate prophylaxis in haemophilia A patients. Haemophilia. 2023 Jan;29(1):156-164. doi: 10.1111/hae.14700. Epub 2022 Nov 21. PMID 36409282